CLINICAL TRIAL: NCT03088891
Title: The Effect of an Increased Intake of Antioxidant-rich Foods on Training Adaptation, Redox-balance and Inflammation Among Elite Athletes During a Moderate Altitude Training Camp
Brief Title: Effect of an Antioxidant-rich Diet During Moderate Altitude Training
Acronym: ALTAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Norwegian School of Sport Sciences (Other); Norwegian Olympic Federation, Oslo, Norway (Unknown)
Responsible Party: Principal Investigator, Rune Blomhoff, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ALTAX
Record Dates: First submitted 2016-09-20; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Oxidative Stress; Adaptation Reaction; Inflammation
Keywords: altitude training; antioxidants; oxidative stress; elite athletes; inflammation; diet
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antioxidant-rich snacks (Experimental): The participants received antioxidant-rich snacks every day during 21 days of moderate altitude training (2300 meters above sea level). The snack included fruits and vegetable smoothies, dark chocolate, walnuts, dried fruits and berries.
  Interventions: Other: Antioxidant-rich snacks
- Control snacks (Placebo Comparator): The participants received antioxidant-depleted snacks every day during 21 days of moderate altitude training (2300 meters above sea level). The snack included milkshake, and other milk-based drinks, biscuits (both sweet and salty), white chocolate.
  Interventions: Other: Control snacks

INTERVENTIONS:
Other: Antioxidant-rich snacks — Bama Smoothies (Bama, Oslo, Norway), Freia Premium Dark Chocolate (Freia, Oslo, Norway), Walnuts (Eldorado, Norway), Dried fruits and berries (Cranberries, Gojiberries, apricots)(Bama, Oslo, Norway and Rema 1000, Norway)
  Arms: Antioxidant-rich snacks
Other: Control snacks — Milkshake (Tine, Oslo, Norway), YT restitusjonsdrikk (Tine, Oslo, Norway), Bixit (Sætre, Oslo, Norway), Ritz (Mondelez, Oslo, Norway), White chololate (Freia, Oslo, Norway)
  Arms: Control snacks

SUMMARY:
Athletes, especially in endurance sports, are at increased risk of oxidative stress and inflammation-related diseases and injuries. The production of reactive oxygen and nitrogen species (RONS) and inflammatory markers increase during exercise and especially during altitude training. Antioxidant supplementation is commonly used among athletes in the belief that it prevents oxidative stress and oxidative damage. A transient increase of RONS is however necessary to activate signaling cascades initiating training adaptation. Antioxidant supplementation has been shown to inhibit the exercise effects in several independent studies, possibly by interfering/reducing the signal cascades initiated by RONS. However, it is unknown whether a high intake of antioxidant rich foods can affect the amount of RONS, inflammation markers and/or training adaptation. The investigators want to examine whether an increased intake of natural antioxidants in the form of antioxidant-rich foods fruits, vegetables and berries, in line with the official Norwegian dietary advice can affect antioxidant status, immune function and training adaptation associated with altitude training in Norwegian elite athletes.

ELIGIBILITY:
Inclusion Criteria:

* National team athletes, summer endurance sports

Exclusion Criteria:

* Allergies in conflict with the intervention foods
* Use of medication that could affect training and performance
* Injuries that could affect training and performance

Ages: 16 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percent change in performance (sport specific tests will be aggregated to one outcome by the use of percent change) | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  Cycling: 10 000 m on a bike roller; Rowing: 2000 meter on Concept2-apparatus; Paddling: 1000 meter Concept2-apparatus; Swimming: 200 meter
Training adaptation | Measured one week before, and one week after the moderate altitude training camp
  change in Vo2-max
Training adaptation for swimmers | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  For swimming only: 100 meter max speed

SECONDARY OUTCOMES:
Change in biomarkers of inflammation | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  change in cytokine profile e.g. IL-6 ,TNF, CRP measured by multiplex technology
change in lean body mass | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  measured by DXA (iDXA; GE Healthcare)
Bone mineral density | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  measured by DXA (iDXA; GE Healthcare)
change in fat mass | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  measured by DXA (iDXA; GE Healthcare)
change in body composition | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  measured by DXA (iDXA; GE Healthcare)
change in body weight | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  measured by standardized scale
Dietary intake (change in food and nutrient intake) | Measured one and three week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  measured by repeated 24 hour recalls
Change in antioxidant status | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  e.g. FRAP, ORAC, dROM, isoprostanes measured by HPLC
biomarkers of antioxidant-rich foods | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  e.g. carotenoids, flavonoids measured by HPLC
Change in whole blood gene expression | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  Fasting blood samples (PAX-tubes) and samples taken after physical stress test (PAX-tubes). RNA will be isolated and gene expression measured
Change in blood lipids | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
Change hormones | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
Change in micronutrients | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  e.g. iron status
change response to stress test | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
Change in hemoglobin | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  CO-rebreathing-method
change in blood volume | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  CO-rebreathing-method
change in plasma volume | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  CO-rebreathing-method
Change in lactate | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
Total training load | Measured one week before, during (in week 1 and 3 of the camp) and one week after the moderate altitude training camp
  Training diary

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - University of Oslo, Oslo
  - Norwegian Olympic Federation, Oslo

REFERENCES:
- [Derived] Koivisto-Mork AE, Paur I, Paulsen G, Garthe I, Raastad T, Bastani NE, Blomhoff R, Bohn SK. Dietary Adjustments to Altitude Training in Elite Endurance Athletes; Impact of a Randomized Clinical Trial With Antioxidant-Rich Foods. Front Sports Act Living. 2020 Aug 26;2:106. doi: 10.3389/fspor.2020.00106. eCollection 2020. PMID 33345095